CLINICAL TRIAL: NCT04229147
Title: Ledderhose Disease - Long Term Effects of Radiotherapy Treatment. LedRad LTE - Study
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: RT2019-09
Record Dates: First submitted 2019-07-05; First posted 2020-01-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Ledderhose Disease
Keywords: Radiotherapy; Pain; Side effect; Satisfaction
MeSH Terms: conditions — Fibromatosis, Plantar; Pain; Personal Satisfaction | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Patients who received a total dose of 30 Gy

SUMMARY:
The aim of the LedRad LTE study is to determine the current complaints, late side effects and satisfaction of patients who were treated with radiotherapy for Ledderhose disease at least two years ago.

ELIGIBILITY:
Patients treated with radiotherapy for Ledderhose disease at the UMCG at least 2 years ago

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Ledderhose disease and treated with radiotherapy at least 2 years ago at the UMCG
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Current pain | at least 2 years after treatment
  Determine pain with the numeric rating scale. A 11-point pain scale ranging from 0=no pain to 10=worst pain

SECONDARY OUTCOMES:
Worst pain | at least 2 years after treatment
  Determine pain with the numeric rating scale. A 11-point pain scale ranging from 0=no pain to 10=worst pain
Quality of Life | at least 2 years after treatment
  Assess the impact on quality of life of the treatment with radiotherapy for this study population with the EURO-Qol-5D-5L
Late side effects of treatment | at least 2 years after treatment
  Is treatment still effective and/or are there any (unknown) side effects of treatment
Satisfaction with radiotherapy treatment for Ledderhose disease | at least 2 years after treatment
  Determine patient satisfaction with the radiotherapy treatment for Ledderhose disease using a self developed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No